CLINICAL TRIAL: NCT04833465
Title: Development of a Therapeutic Endpoint in Pediatric Rheumatologic Conditions
Status: Recruiting | Type: Observational
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Julia Finkel, Professor of Anesthesiology and Pediatrics, Children's National Research Institute
Other Study IDs: Pro00015629
Record Dates: First submitted 2021-04-02; First posted 2021-04-06 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Juvenile Idiopathic Arthritis; Systemic Lupus Erythematosus; Fibromyalgia
MeSH Terms: conditions — Arthritis, Juvenile; Lupus Erythematosus, Systemic; Fibromyalgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- JIA: Patients ages 5-21 with a diagnosis of JIA.
  Interventions: Other: No Intervention
- SLE: Patients ages 5-21 with a diagnosis of SLE.
  Interventions: Other: No Intervention
- FM: Patients ages 5-21 with a diagnosis of FM.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
The overarching goal of this study is the development of a physiologic endpoint of pain and treatment effect in three distinct rheumatology populations. This would enable objective assessment of pain and treatment in these populations and enable a much more precise approach to treatment. Such an endpoint stands to significantly improve outcomes in these patients by eliminating the need for a trial-and-error approach to treatment. This is a single site observational study that aims to collect initial pilot data in three distinct patient groups. As this is observational, there is no randomization or blinding in the study. Patients will be followed for a period of one year after enrollment. Baseline measurements will be taken at the time of enrollment, and at each subsequent standard of care clinic visit as feasible, for a period of one year. As this is an observational study, there will be no change to the treatment for any patient due to research activities. The primary objective of this study is the characterization of the nociceptive index in three pediatric rheumatology populations. The secondary objective is the characterization of the nociceptive index in these populations in response to standard of care interventions. This is necessary to demonstrate the ability of this approach to serve as an endpoint of treatment effect.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible for inclusion in the study, an individual must meet all of the following criteria:

* Male or female ≥ 5 years of age at screening.
* Documentation of a JIA, SLE or FM diagnosis as evidenced by history

Exclusion Criteria:

Any individual who meets any of the following criteria will be excluded from participation in this study:

• Documented history of eye disease precluding pupillometry

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 30 subjects from each of the three populations of interest will be enrolled for this study.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2021-07-16 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Index Characterization | 1 Year
  The primary objective of this study is the characterization of the nociceptive index in three pediatric rheumatology populations.

SECONDARY OUTCOMES:
Treatment Effect | 1 Year
  The secondary objective is the characterization of the nociceptive index in these populations in response to standard of care interventions. This is necessary to demonstrate the ability of this approach to serve as an endpoint of treatment effect.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's National Health System, Washington D.C., District of Columbia, United States